CLINICAL TRIAL: NCT04147169
Title: Compassionate End of Life Care in the ICU: Evaluating the Value, Transferability, Affordability, and Sustainability and Value of the 3 Wishes Project
Brief Title: A Multicenter Implementation Study of the 3 Wishes Project
Acronym: 3WP
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: The Greenwall Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3WP_Multicenter
Record Dates: First submitted 2019-10-08; First posted 2019-10-31 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Death; Communication, Multidisciplinary; Empathy; Compassion; Family Members; Bereavement; Empowerment; Patient Engagement
Keywords: Compassionate; End-of-Life Care; Interpersonal connections
MeSH Terms: conditions — Death; Communication; Empowerment; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dying patients: Dying patients admitted to the Intensive Care Unit who are approaching end-of-life.
  Interventions: Behavioral: Focused end-of-life conversations to promote connections among patients, family members and clinicians.

INTERVENTIONS:
Behavioral: Focused end-of-life conversations to promote connections among patients, family members and clinicians. — All eligible patients and families who were invited to participate in wish elicitation and implementation. For family interviews, criterion sampling was used. For the clinician focus groups, criterion sampling was used, based on involvement in the care of a 3WP patient. For the manager/hospital administrator interviews, purposive sampling was used, based on relevant leadership positions. Investigators employed qualitative and quantitative methods to collect and analyze data. Quantitative data include characteristics of patients, families and clinicians, questionnaire responses from families who agree to interviews, and clinicians who agree to focus groups, respectively, types of wishes elicited and implemented, and their cost. Qualitative data was obtained through individual family interviews, inter-professional clinician focus groups, project team field notes, additional ideas about the costs and benefits of the project from manager interviews, and analysis of project documents.

SUMMARY:
The 3 Wishes Project (3WP) was created to promote the connections between patients, family members, and clinicians that are foundational to empathic end-of-life care. It provides a scaffold for discussions about preferences and values at the end of life and leads to acts of compassion that arise from soliciting and implementing wishes that honour the dying patient. In a single center, investigators previously reported how the 3 Wishes Project forges interpersonal connections among patients, family members and clinicians, eases family grief, and offers experiential end of life education for clinicians-in-training.

The objective of this study was to evaluate whether the 3 Wishes Project could enhance compassionate care for dying patients and their families when implemented as a multicenter program. Given the importance of empowering frontline staff to adapt the 3WP to their own practice patterns, investigators did not protocolize this approach to personalizing end-of-life care. Investigators conceptualized this study as a formative evaluation of 3WP to examine its 1) Value: as experienced by family members, frontline clinicians, ICU managers and hospital administrators; 2) Transferability: successful implementation beyond the original ICU by a different mix of clinicians; 3) Affordability: cost of wishes being less than $50/patient; 4) Sustainability: project continuation beyond the first year of evaluation.

DETAILED DESCRIPTION:
This is a mixed-methods formative program evaluation of the 3 Wishes Project implemented in ICUs in Toronto, Vancouver, Los Angeles, and the original center in Hamilton.

Implementation of the 3WP was aligned with the interests and cultural norms at each center, adapted by local clinicians with the resources available, assisted by close contact and informational guidance from the original site. Each center implemented the 3WP as both a clinical program and research project. Participating ICUs were all located in academic tertiary care centers with some differing features.

Design: This is a multi-center mixed-methods implementation and formative evaluation study. Data collection will be quantitative and qualitative (interviews and focus groups). Investigators will take a systems-level approach to produce information on how to implement the 3 Wishes Project in different settings, each with its own social microcosm, affordances and constraints.

Specific Aims are: 1) For patients, to provide compassionate end of life care consistent with their values and preferences; 2) For family members, to evaluate the project's impact on family views on end of life care; 3) For clinicians, to explore the project's impact on compassion, resilience, moral distress, and views on end of life care; 4) For ICU managers, to learn of any barriers to implementation and strategies for facilitation; and 5) For hospital administrators, to understand perceived costs and institutional benefits such as alignment with priorities for end of life care.

Investigators will use a case study approach examining particularities of the 'eco-system' of each ICU to examine how the 3 Wishes Project operates in each setting. This examination will include the constraints, affordances, and impacts available from the staffing model, organizational culture, end of life policies and administrative structure. An understanding of each ICU will be developed, with comparisons made to illuminate broader findings and suggest strategies for expanding the project elsewhere.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patient is >18 years of age (a subgroup analysis will be conducted on those >65 years of age);
2. Patient has a >95% of dying during the ICU stay as judged by the ICU attending physician; or
3. a decision has been made to withdraw or withhold advanced life support in anticipation of death.

Patient/Family Exclusion Criteria:

1. Prohibitive communication challenges (e.g., serious psychological or psychiatric illness in the patient and/or family, inability of patient and/or family to communicate reasonably well in English or other language for which an interpreter exists - professional staff or otherwise);
2. Prohibitive logistics (e.g., patient admitted to the ICU for <24 hours, or anticipated to die within 24 hours of screening)
3. Patient or family declines. (Note that a patient who has "no family" (even very broadly defined as friends and neighbours, or community members and case workers for homeless persons) would not be excluded from the wish elicitation and implementation component of the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be admitted into the Intensive Care Unit, who are critically ill and have a poor outcome (likely to die during the ICU admission). When death looms in the ICU, people invariably interpret life through a lens of meaning - existential, spiritual, and relational. Through this lens, the 3 Wishes Project clearly facilitates holistic care, beyond the physical, to honour and celebrate a life. Staff are empowered and encouraged to sensitively elicit and then implementing at least 3 wishes from patients, family members, and/or clinicians caring for dying patients.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Perceptions and beliefs about value of the program | Through study completion, an average of 1 year.
  Given the nascent knowledge of experiences and perceptions of value, it is important that investigators first understand which program elements family members and clinicians appreciate, and what their experiences of these elements are. In future research, investigators will then measure achievement in those domains. Accordingly, in this study investigators will solicit open-ended, qualitative perceptions of value of the program from family members, clinicians, and ICU managers and hospital administrators. This information will be analyzed inductively to generate domains of value which may be measured in future research. Inductive analysis involves generation of categories and domains directly from the data, without pre-conceived notions of what these categories or domains might be. By generating understanding of the types of value family members, clinicians and managers see in this program, investigators will be able to devise ways to measure this value in future research.
Transferability as indicated by successful establishment in 3 new ICU settings | Through study completion, an average of 1 year.
  Successful implementation beyond the original ICU by a different mix of clinicians.
Affordability: cost of wishes being less than $50/patient. | Through study completion, an average of 1 year
  The $50/patient figure quoted does not refer to patient compensation. Instead, it refers to the cost of running the intervention for each enrolled patient. Given the individually-adapted nature of this intervention, the costs will vary per participant. Affordability of the program to the ICU running the program is an essential part of information collected in this program evaluation.
  Affordability will be informed by mean cost per wish and per patient at each center and overall. Also, investigators will perform a cost description of the project including both direct and indirect costs.
Sustainability of the intervention after the research study has been completed. | 6 months after study completion
  Sustainability will be affirmed if the project remains operational in each ICU in July 2019.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Participants did not agree to data sharing (qualitative or quantitative). Also, in some instances, this would be identifying. Feel free to contact us for further information.

REFERENCES:
- [Derived] Vanstone M, Neville TH, Swinton ME, Sadik M, Clarke FJ, LeBlanc A, Tam B, Takaoka A, Hoad N, Hancock J, McMullen S, Reeve B, Dechert W, Smith OM, Sandhu G, Lockington J, Cook DJ. Expanding the 3 Wishes Project for compassionate end-of-life care: a qualitative evaluation of local adaptations. BMC Palliat Care. 2020 Jun 30;19(1):93. doi: 10.1186/s12904-020-00601-5. PMID 32605623
- [Derived] Vanstone M, Neville TH, Clarke FJ, Swinton M, Sadik M, Takaoka A, Smith O, Baker AJ, LeBlanc A, Foster D, Dhingra V, Phung P, Xu XS, Kao Y, Heels-Ansdell D, Tam B, Toledo F, Boyle A, Cook DJ. Compassionate End-of-Life Care: Mixed-Methods Multisite Evaluation of the 3 Wishes Project. Ann Intern Med. 2020 Jan 7;172(1):1-11. doi: 10.7326/M19-2438. Epub 2019 Nov 12. PMID 31711111